CLINICAL TRIAL: NCT00201253
Title: Expression of Tuberculosis in the Lung
Status: Completed | Type: Observational
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 286; R01HL051630 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cell culture supernatants and cell lysates from bronchoalveolar cells, as well as peripheral blood mononuclear cells.
  Bronchoalveolar lavage fluid

INTERVENTIONS:
Other: Bronchoalveolar lavages and venipunctures only

SUMMARY:
The purpose of this study is to assess lung immune responses in patients with active pulmonary tuberculosis (TB) and in healthy control persons who are exposed to Mycobacterium tuberculosis in households of patients with TB or who are unexposed.

DETAILED DESCRIPTION:
BACKGROUND:

M. tuberculosis infects a third of the world's population, and TB is the leading cause of morbidity and mortality due to a single infectious agent. However, only 5% to 10% of M. tuberculosis-infected subjects without an underlying immunodeficiency develop disease during their lifetimes. Therefore protective immunity is induced in the majority of subjects. Understanding correlates of protection against M. tuberculosis in humans is needed to better direct efforts in the development of antituberculosis vaccines.

DESIGN NARRATIVE:

Patients are treated according to good clinical practice; however, no study medications are given as part of the research study. This study involves a one-time bronchoalveolar lavage and venipuncture to obtain immune cells for laboratory studies of immune responses.

ELIGIBILITY:
Inclusion Criteria:

* TB patients who are 18 to 65 years old
* Clinical and radiographic signs and symptoms consistent with pulmonary TB
* Start date of antituberculous chemotherapy less than 10 days prior to procedures
* Sputum smear positive for acid fast bacilli
* Drug-sensitive, culture-confirmed growth of M. tuberculosis from sputum
* Willing to provide informed consent for participation in bronchoalveolar lavage and venipuncture studies

Exclusion Criteria:

* TB patients who have HIV-1 coinfection
* History of any chronic medical condition requiring daily medication (including diabetes mellitus, hypertension, chronic infections, renal or cardiac failure, and peptic ulcer disease)
* History of asthma or upper or lower respiratory tract infection within 2 months of the study
* Hemoglobin level less than 10g/dl

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tuberculosis and household contacts of patients with tuberculosis.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2000-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pulmonary immune responses associated with resistance and susceptibility to Mycobacterium tuberculosis infection (measured at baseline) | one week

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Ellner, Principal Investigator — UMDNJ-New Jersey Medical School
Locations (2):
- UMDNJ-New Jersey Medical School, Newark, New Jersey, United States
- Instituto Nacional de Enfermedades Respiratorias (INER), Mexico City, Mexico

REFERENCES:
- [Background] Rivas-Santiago B, Schwander SK, Sarabia C, Diamond G, Klein-Patel ME, Hernandez-Pando R, Ellner JJ, Sada E. Human beta-defensin 2 is expressed and associated with Mycobacterium tuberculosis during infection of human alveolar epithelial cells. Infect Immun. 2005 Aug;73(8):4505-11. doi: 10.1128/IAI.73.8.4505-4511.2005. PMID 16040961